CLINICAL TRIAL: NCT06512168
Title: Measuring Aided Language Development
Acronym: MALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of New Mexico (Other); University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Jennifer Kent-Walsh, Pegasus Professor & Associate Dean of Research, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AWD00006137; 1R01DC021160-01A1 (NIH)
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome; Cerebral Palsy; Apraxia of Speech; Speech Sound Disorder; Speech Disorders in Children; Speech and Language Disorder
Keywords: Augmentative and Alternative Communication; Complex Communication Needs; Assistive Technology; AAC
MeSH Terms: conditions — Down Syndrome; Cerebral Palsy; Apraxias; Speech Sound Disorder; Speech; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): AAC Generative Language Intervention
  Interventions: Behavioral: AAC Generative Language Intervention

INTERVENTIONS:
Behavioral: AAC Generative Language Intervention — Aided AAC Language Input/Output Intervention

SUMMARY:
The focus of the current study is to systematically investigate the psychometric properties of a range of aided language measures, which are based on the Graphic Symbol Utterance and Sentence Development Framework (Binger & Kent-Walsh).

DETAILED DESCRIPTION:
Our central hypotheses are: (1) psychometrically sound measures can be established to capture growth within and across different dimensions of language acquisition, and (2) some elicitation contexts will be better than others at capturing aided language growth. Specific Aim 1 identifies valid measures to characterize aided language progress. Aim 1A uses existing data to document the psychometric properties of a range of aided language measures for preschoolers at the early stages of aided communication acquisition who have received 4 months of aided language intervention. Aim 1B analyzes language progression for high-performing aided communicators who will receive 24 months of intervention; this allows for investigation across all phases of early aided language acquisition. Specific Aim 2 identifies elicitation contexts that demonstrate the most productive aided language use. Achievement of the aims will result in measures that demonstrate strong reliability, differentiate growth for different populations, describe different dimensions of language growth, and are clinically feasible.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Identification of Down Syndrome or Cerebral Palsy + Significant Speech Impairment
* Must Speak English as a Primary Language
* Must Be Able to Express At Least 25 Words (using any communication mode)
* Must Be Able to Accurately Select Picture Symbols on iPad Communication App with at Least 50% Accuracy
* Vision and Hearing within Functional Limits or Corrected to be within Functional Limits for Study Activities

Exclusion Criteria:

* Clinical Diagnosis of Autism or Social Communication Disorder
* Primary Language Spoken is A Language Other than English

Ages: 42 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Aided AAC Utterance Length | 24 Months
  Aided AAC Sentence Length Measured in Morphemes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida - Innovative Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
NICHD Data and Specimen Hub